CLINICAL TRIAL: NCT05265065
Title: A Randomised Controlled Trial to Assess the Immunogenicity, Safety and Reactogenicity of Standard Dose Versus Fractional Doses of COVID-19 Vaccine (Pfizer-BioNTech) Given as a Booster Dose After Priming With Sinopharm, AstraZeneca or Sputnik in Healthy Adults in Mongolia
Brief Title: Evaluation of Full Versus Fractional Dose of COVID-19 Vaccine Given as a Booster for the Prevention of COVID-19 in Adults in Mongolia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); The Peter Doherty Institute for Infection and Immunity (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 81800
Record Dates: First submitted 2022-03-01; First posted 2022-03-03 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
Keywords: Booster dose; Pfizer; fractional and standard doses; COVID-19 vaccination; mRNA vaccine
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Intervention Model Description: Study participants who have received two doses of either Sinopharm, AstraZeneca or Sputnik vaccine as their primary vaccine will be randomised into one of two groups. The two groups consist of a standard or fractional dose of Pfizer vaccine.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants and those evaluating reactogenicity will be blinded to the vaccine allocation for the first 28 days following vaccination. After that, both clinical investigators and participants will be aware of their investigational product allocation. Laboratory staff will remain blinded to the investigational product allocation during the immunology testing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard Pfizer-BioNTech booster group (Active Comparator): Biological/Vaccine: Tozinameran - Standard Dose
  Other Names:
  BNT162b2 Comirnaty Pfizer Covid-19 vaccine
  Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 30 µg in 0.3 ml. Liquid for injection. Single dose.
  Interventions: Biological: Tozinameran - Standard Dose
- Fractional Pfizer-BioNTech booster group (Experimental): Biological/Vaccine: Tozinameran - Standard Dose
  Other Names:
  BNT162b2 Comirnaty Pfizer Covid-19 vaccine
  Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.3 ml. Liquid for injection. Single dose.
  Interventions: Biological: Tozinameran - Fractional Dose

INTERVENTIONS:
Biological: Tozinameran - Standard Dose — Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 30 µg in 0.3 ml. Liquid for injection. Single dose.
  Other Names: BNT162b2; Comirnaty; Pfizer Covid-19 vaccine
  Arms: Standard Pfizer-BioNTech booster group
Biological: Tozinameran - Fractional Dose — Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.15 ml. Liquid for injection. Single dose.
  Other Names: BNT162b2; Comirnaty; Pfizer Covid-19 vaccine
  Arms: Fractional Pfizer-BioNTech booster group

SUMMARY:
This clinical trial is a single-blind, randomised study to determine the reactogenicity and immunogenicity of severe acute respiratory syndrome-coronavirus-2 (SARS-CoV-2) vaccine (Pfizer-BioNTech) as booster dose in adults, who have previously received either Sinopharm (BBIBP-CorV®), AstraZeneca (ChAdOx1-S, or Vaxzevria®) or Sputnik V (Gam-COVID-Vac®) as their primary doses 6 to 9 months earlier. Both standard and fractional doses will be tested.

Participants are healthy adults aged 18 years or older, with no upper age limit. Procedures will be implemented to ensure participants of all ages (aged 18 and above) are included and that there is an even age distribution (<50 and ≥50 years) in each group. There will be a total of 6 groups (Sinopharm-standard dose Pfizer, Sinopharm-fractional dose Pfizer, AstraZeneca-standard dose Pfizer, AstraZeneca-fractional dose Pfizer, Sputnik - standard dose Pfizer, Sputnik - fractional dose Pfizer), with 200 participants per group for Sinopharm and 100 for AstraZeneca and Sputnik.

DETAILED DESCRIPTION:
As per brief summary

ELIGIBILITY:
Inclusion Criteria:

1. Have completed two doses of Sinopharm, AstraZeneca or Sputnik vaccines with the recommended schedule 6 months prior to the date of enrolment
2. Willing and able to give written informed consent
3. Aged 18 years or above
4. Willing to complete the follow-up requirements of the study

Exclusion Criteria:

1. Received 3 doses of COVID-19 vaccine
2. Received 2 doses of COVID-19 less than 6 months prior to the start of the trial
3. Currently on immunosuppressive medication or anti-cancer chemotherapy
4. HIV infection
5. Congenital immune deficiency syndrome
6. Has received immunoglobulin or other blood products in the 3 months prior to vaccination
7. Study staff and their relatives
8. Have a history of a severe allergic reaction to any COVID-19 vaccines or have a medical exception to receiving further COVID-19 vaccines

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2024-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tsetsegsaikhan Batmunkh, MD, Principal Investigator — Ministry of Health, Mongolia; Kim Mulholland, MD/Prof, Principal Investigator — Murdoch Childrens Research Institute
Locations (1):
- District Health Centre, Ulaanbaatar, Mongolia

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data to ethically approved studies in cases where participants have indicated on the consent form that they consent to the use of their data and where consistent with terms of collaboration agreements.
Supporting Information: Study Protocol, ICF
Time Frame: Individual participant data (IPD) sharing plans in development
Access Criteria: IPD sharing plans in development
URL: https://www.melbournechildrens.com/mctc/

REFERENCES:
- [Background] Munro APS, Janani L, Cornelius V, Aley PK, Babbage G, Baxter D, Bula M, Cathie K, Chatterjee K, Dodd K, Enever Y, Gokani K, Goodman AL, Green CA, Harndahl L, Haughney J, Hicks A, van der Klaauw AA, Kwok J, Lambe T, Libri V, Llewelyn MJ, McGregor AC, Minassian AM, Moore P, Mughal M, Mujadidi YF, Murira J, Osanlou O, Osanlou R, Owens DR, Pacurar M, Palfreeman A, Pan D, Rampling T, Regan K, Saich S, Salkeld J, Saralaya D, Sharma S, Sheridan R, Sturdy A, Thomson EC, Todd S, Twelves C, Read RC, Charlton S, Hallis B, Ramsay M, Andrews N, Nguyen-Van-Tam JS, Snape MD, Liu X, Faust SN; COV-BOOST study group. Safety and immunogenicity of seven COVID-19 vaccines as a third dose (booster) following two doses of ChAdOx1 nCov-19 or BNT162b2 in the UK (COV-BOOST): a blinded, multicentre, randomised, controlled, phase 2 trial. Lancet. 2021 Dec 18;398(10318):2258-2276. doi: 10.1016/S0140-6736(21)02717-3. Epub 2021 Dec 2. PMID 34863358
- [Derived] Batmunkh T, Neal EFG, Amraa O, Mazarakis N, Altangerel B, Avaa N, Batbayar L, Batsukh K, Bright K, Burentogtokh T, Do LAH, Dorj G, Hart JD, Jamiyandorj O, Javkhlantugs K, Jigjidsuren S, Justice F, Li S, Mashbaatar K, Moore KA, Namjil N, Nguyen CD, Ochirbat B, Surenjav U, Thomson H, Tsolmon B, Licciardi PV, von Mollendorf C, Mulholland K. Immunogenicity and safety at twelve months of fractional and standard BNT162b2 booster doses in adults primed with ChAdOx1-S, BBIBP-CorV, or Gam-COVID-Vac in Mongolia: a randomised controlled trial. Vaccine. 2025 Nov 14;66:127840. doi: 10.1016/j.vaccine.2025.127840. Epub 2025 Oct 9. PMID 41072276
- [Derived] Batmunkh T, Moore KA, Thomson H, Altangerel B, Amraa O, Avaa N, Batbayar L, Batsukh K, Bright K, Burentogtokh T, Ha Do LA, Dorj G, Hart JD, Javkhlantugs K, Jigjidsuren S, Justice F, Li S, Licciardi PV, Mashbaatar K, Mazarakis N, Neal EFG, Nguyen CD, Ochirbat B, Tsolmon B, Tuya A, Surenjav U, von Mollendorf C, Mulholland K. Immunogenicity, safety, and reactogenicity of a half- versus full-dose BNT162b2 (Pfizer-BioNTech) booster following a two-dose ChAdOx1 nCoV-19, BBIBP-CorV, or Gam-COVID-Vac priming schedule in Mongolia: a randomised, controlled, non-inferiority trial. Lancet Reg Health West Pac. 2023 Nov 21;42:100953. doi: 10.1016/j.lanwpc.2023.100953. eCollection 2024 Jan. PMID 38357398
- See also: Quarter-dose of Moderna COVID vaccine still rouses a big immune response — https://www.nature.com/articles/d41586-021-01893-0
- See also: US Food and Drug Administration (FDA). Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials 2007 — https://www.fda.gov/media/73679/download

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There are two study arms (i.e. groups to which participants were randomised), as per "Arms and Interventions" in Protocol Section, corresponding to the primary analysis comparing a full dose to a fractional dose. Stratified randomisation was performed to ensure balanced randomisation according to the primary vaccine received (prior to this study) and age for secondary subgroup analyses. The Participant Flow was edited to reflect the randomisation of participants into two arms.
Groups:
- Standard: 30µg Pfizer-BioNTech booster dose
- Fractional: 15µg Pfizer-BioNTech booster dose
Period: Overall Study
Arm/Group | Standard | Fractional
Started | 300 | 301
Received Allocated d Dose | 299 (1 withdrew prior to receiving study vaccine) | 299 (2 withdrew prior to receiving study vaccine)
Included in Day 28 Immunogenicity Analysis | 292 (7 missed Day-28 visit) | 295 (4 missed Day-28 visit)
Completed (Included in Month-12 immunogenicity analysis) | 282 | 285
Not Completed | 18 | 16

BASELINE CHARACTERISTICS:
Groups:
- AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Standard Pfizer-BioNTech Booster Group: Previously received two doses of AstraZeneca as primary COVID-19 vaccine
  Tozinameran - Standard Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 30 µg in 0.3 ml. Liquid for injection. Single dose.
- AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Fractional Pfizer-BioNTech Booster Group: Previously received two doses of AstraZeneca as primary COVID-19 vaccine
  .
  Tozinameran - Fractional Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.15 ml. Liquid for injection. Single dose.
- Sinopharm (BBIBP-CorV®)- Standard Pfizer-BioNTech Booster Group: Previously received two doses of Sinopharm as primary COVID-19 vaccine
  Tozinameran - Standard Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 30 µg in 0.3 ml. Liquid for injection. Single dose.
- Sinopharm (BBIBP-CorV®)- Fractional Pfizer-BioNTech Booster Group: Previously received two doses of Sinopharm as primary COVID-19 vaccine
  Tozinameran - Fractional Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.15 ml. Liquid for injection. Single dose.
- Sputnik V (Gam-COVID-Vac®)- Standard Pfizer-BioNTech Booster Group: Previously received two doses of Sputnik as primary COVID-19 vaccine
  Tozinameran - Standard Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 30 µg in 0.3 ml. Liquid for injection. Single dose.
- Sputnik V (Gam-COVID-Vac®)- Fractional Pfizer-BioNTech Booster Group: Previously received two doses of Sputnik as primary COVID-19 vaccine
  Tozinameran - Fractional Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.15 ml. Liquid for injection. Single dose.
- Total: Total of all reporting groups
Arm/Group | AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Standard Pfizer-BioNTech Booster Group | AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Fractional Pfizer-BioNTech Booster Group | Sinopharm (BBIBP-CorV®)- Standard Pfizer-BioNTech Booster Group | Sinopharm (BBIBP-CorV®)- Fractional Pfizer-BioNTech Booster Group | Sputnik V (Gam-COVID-Vac®)- Standard Pfizer-BioNTech Booster Group | Sputnik V (Gam-COVID-Vac®)- Fractional Pfizer-BioNTech Booster Group | Total
Number analyzed (Participants) | 65 | 65 | 201 | 200 | 34 | 36 | 601
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 3 | 0 | 0 | 0 | 3
  Between 18 and 65 years | 65 | 65 | 189 | 186 | 30 | 35 | 570
  >=65 years | 0 | 0 | 9 | 14 | 4 | 1 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.5 [32.2 to 45.8] | 40.2 [33.7 to 49.6] | 47.8 [31.4 to 57.7] | 48.8 [32 to 56.9] | 43.1 [32.1 to 52.7] | 41.3 [34.7 to 50.3] | 44 [32.4 to 54.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 32 | 115 | 114 | 19 | 14 | 327
  Male | 32 | 33 | 86 | 86 | 15 | 22 | 274
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Mongolia | 65 | 65 | 201 | 200 | 34 | 36 | 601
BMI [Number; unit: kg/m2] | 26.3 | 25.4 | 24.6 | 24.8 | 25.3 | 25.8 | 25.2

OUTCOME MEASURES:

1. Primary Outcome: Seroresponse
Description: Serum samples collected at 28-days post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific IgG antibodies using IgG ELISA. The primary endpoint is the seroresponse rate at the Day-28 visit. The seroresponse rate at the individual level is defined as either a ≥4-fold rise in binding antibodies at the Day-28 visit compared to baseline (pre-vaccination) with a titre of <200 BAU/ml, a ≥2-fold rise among participants with a baseline (pre-vaccination) titre of >200 BAU/ml, or a ≥4-times the lower limit of detection if baseline levels are lower than the limit of detection.
Time Frame: 28-days post booster vaccination
Population: The analysis of immunogenicity endpoints included all participants with outcome data.
  There are two study arms, as per "Arms and Interventions" in Protocol Section, corresponding to the primary analysis comparing a full dose to a fractional dose. Stratified randomisation was performed to ensure balanced randomisation according to the primary vaccine received (prior to this study) and age for secondary subgroup analyses. The primary outcome is unstratified.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Fractional
Number analyzed (Participants) | 292 | 295
Participants | 253 | 250
Statistical Analysis 1: Comparison: Standard vs Fractional; Non-inferiority margin of -10% (absolute difference) and a one-sided significance level of 5%; Test type: Non-Inferiority — Non-inferiority margin of -10% (absolute difference) and a one-sided significance level of 5%. The sample size calculation assumed an estimated seroresponse rate of 95% in both half- and full-dose arms, a non- inferiority margin of -10% (absolute difference), a one-sided significance level of5%, and no loss to follow- up. Under this scenario, a sample size of 100 per arm provides 90% power to compare seroresponse rates between arms under the non-inferiority framework; Regression, Logistic; Risk Difference (RD) = -2.9, 95% CI 2-sided [-7.7 to 2.0] — The difference in seroresponse was adjusted for age group, priming vaccine, duration between first and second dose, duration between second and third (study) dose, study day of blood draw, and baseline anti-spike IgG (IgG)

2. Primary Outcome: Solicited Grade 3 or 4 Local or Systemic Reaction
Description: Questionnaire to document solicited reactions is developed specifically for this study. Data will be reported as the proportion of participants who report grade 3 or 4 reactions by each intervention arm. Solicited reactions such as pain, tenderness, erythema/redness, induration, swelling, fever, nausea, vomiting, headache, fatigue/malaise, myalgia, arthralgia, diarrhea, enlarged lymph nodes will be collected from the participants 7 days post-vaccination.
Time Frame: 7 days post booster vaccination
Population: The reactogenicity and safety analysis populations included all randomised participants who received a study vaccine, according to the vaccine received.
  There are two study arms, as per "Arms and Interventions" in Protocol Section. Stratified randomisation was performed to ensure balanced randomisation according to the primary vaccine received (prior to this study) and age for secondary subgroup analyses. The primary outcome is unstratified.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard | Fractional
Number analyzed (Participants) | 299 | 299
Participants | 6 | 4

3. Secondary Outcome: Seroresponse by Priming Vaccine Strata
Description: Serum samples collected at 28-days post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific IgG antibodies using IgG ELISA. The primary endpoint is the seroresponse rate at the Day-28 visit. The seroresponse rate at the individual level is defined as either a ≥4-fold rise in binding antibodies at the Day-28 visit compared to baseline (pre-vaccination) with a titre of <200 BAU/ml, a ≥2-fold rise among participants with a baseline (pre-vaccination) titre of >200 BAU/ml, or a ≥4-times the lower limit of detection if baseline levels are lower than the limit of detection.
  Priming strata (previously COVID vaccination): AstraZeneca (ChAdOx1-S, or Vaxzevria®); Sinopharm (BBIBP-CorV®); Sputnik V (Gam-COVID-Vac®)
Time Frame: 28-days post booster vaccination
Population: The analysis of immunogenicity endpoints included all participants with outcome data
Measure: Count of Participants; unit: Participants
Arm/Group | AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Standard Pfizer-BioNTech Booster Group | AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Fractional Pfizer-BioNTech Booster Group | Sinopharm (BBIBP-CorV®)- Standard Pfizer-BioNTech Booster Group | Sinopharm (BBIBP-CorV®)- Fractional Pfizer-BioNTech Booster Group | Sputnik V (Gam-COVID-Vac®)- Standard Pfizer-BioNTech Booster Group | Sputnik V (Gam-COVID-Vac®)- Fractional Pfizer-BioNTech Booster Group
Number analyzed (Participants) | 65 | 62 | 194 | 198 | 33 | 35
Participants | 55 | 52 | 170 | 169 | 28 | 29
Statistical Analysis 1: Comparison: AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Standard Pfizer-BioNTech Booster Group vs AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Fractional Pfizer-BioNTech Booster Group; Test type: Non-Inferiority — Non-inferiority margin of -10% (absolute difference); Regression, Logistic; Risk Difference (RD) = -2.4, 95% CI 2-sided [-16.1 to 11.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Sinopharm (BBIBP-CorV®)- Standard Pfizer-BioNTech Booster Group vs Sinopharm (BBIBP-CorV®)- Fractional Pfizer-BioNTech Booster Group; Test type: Non-Inferiority — Non-inferiority margin of -10% (absolute difference); Regression, Logistic; Risk Difference (RD) = -3.1, 95% CI 2-sided [-9.5 to 3.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Sputnik V (Gam-COVID-Vac®)- Standard Pfizer-BioNTech Booster Group vs Sputnik V (Gam-COVID-Vac®)- Fractional Pfizer-BioNTech Booster Group; Test type: Non-Inferiority — Non-inferiority margin of -10% (absolute difference); Regression, Logistic; Risk Difference (RD) = -0.5, 95% CI 2-sided [-17.1 to 16.1] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: SARS-CoV-2 Specific IgG Antibodies at Day-28
Description: Serum samples collected at 28-days post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific IgG antibodies using IgG ELISA.
Time Frame: 28-days post booster vaccination
Population: The analysis of immunogenicity endpoints included all participants with outcome data.
Measure: Geometric Mean (95% Confidence Interval); unit: BAU/ml
Arm/Group | Standard | Fractional
Number analyzed (Participants) | 292 | 295
BAU/ml | 4946 [4614 to 5302] | 4619 [4292 to 4970]
Statistical Analysis 1: Comparison: Standard vs Fractional; Test type: Superiority; p = 0.228, Regression, Linear; Geometric Mean Ratio = 0.94, 95% CI 2-sided [0.86 to 1.04] — Adjusted for age group, priming vaccine, duration between 1st and 2nd dose, duration between 2nd and 3rd (study) dose, study day of blood draw, and baseline anti-spike IgG (IgG)

5. Secondary Outcome: SARS-CoV-2 Specific IgG Antibodies at Day-28 by Priming Vaccine Strata
Description: Serum samples collected at 28-days post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific IgG antibodies using IgG ELISA.
  Priming strata (previously COVID vaccination): AstraZeneca (ChAdOx1-S, or Vaxzevria®); Sinopharm (BBIBP-CorV®); Sputnik V (Gam-COVID-Vac®)
Time Frame: 28-days post booster vaccination
Population: The analysis of immunogenicity endpoints included all participants with outcome data
Measure: Geometric Mean (95% Confidence Interval); unit: BAU/ml
Arm/Group | AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Standard Pfizer-BioNTech Booster Group | AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Fractional Pfizer-BioNTech Booster Group | Sinopharm (BBIBP-CorV®)- Standard Pfizer-BioNTech Booster Group | Sinopharm (BBIBP-CorV®)- Fractional Pfizer-BioNTech Booster Group | Sputnik V (Gam-COVID-Vac®)- Standard Pfizer-BioNTech Booster Group | Sputnik V (Gam-COVID-Vac®)- Fractional Pfizer-BioNTech Booster Group
Number analyzed (Participants) | 65 | 62 | 194 | 198 | 33 | 35
BAU/ml | 4394 [3863 to 4997] | 4167 [3550 to 4892] | 5109 [4678 to 5580] | 4970 [4541 to 5438] | 5160 [4128 to 6450] | 3662 [3016 to 4447]
Statistical Analysis 1: Comparison: AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Standard Pfizer-BioNTech Booster Group vs AstraZeneca (ChAdOx1-S, or Vaxzevria®) - Fractional Pfizer-BioNTech Booster Group; Test type: Superiority; p = 0.537, Regression, Linear; Geometric Mean Ratio = 0.94, 95% CI 2-sided [0.77 to 1.15] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Sinopharm (BBIBP-CorV®)- Standard Pfizer-BioNTech Booster Group vs Sinopharm (BBIBP-CorV®)- Fractional Pfizer-BioNTech Booster Group; Test type: Superiority; p = 0.922, Regression, Linear; Geometric Mean Ratio = 0.99, 95% CI 2-sided [0.89 to 1.11] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Sputnik V (Gam-COVID-Vac®)- Standard Pfizer-BioNTech Booster Group vs Sputnik V (Gam-COVID-Vac®)- Fractional Pfizer-BioNTech Booster Group; Test type: Superiority; p = 0.014, Regression, Linear; Geometric Mean Ratio = 0.71, 95% CI 2-sided [0.54 to 0.93] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: SARS-CoV-2 Specific IgG Antibodies at Baseline (Pre Booster), 28- Days, 6- and 12-months Post Booster Vaccination.
Description: Serum samples collected at baseline (pre booster), 28 days, 6- and 12-months post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific IgG antibodies using IgG CMIA. Data will be reported as binding antibody units (BAU)/mL and presented as geometric mean concentration (GMC) and 95% confidence intervals (CI).
Time Frame: Baseline (pre booster), 28 days, 6- and 12-months post booster vaccination
Reporting Status: Not Posted

7. Secondary Outcome: SARS-CoV-2 Specific Neutralising Antibodies at Baseline (Pre Booster), 28 Days-, 6- and 12-months Post Booster Vaccination Measured by Surrogate Virus Neutralization Test (sVNT).
Description: Serum samples collected at baseline (pre booster), 28 days-, 6- and 12-months post booster vaccination from all groups will be evaluated for SARS-CoV-2 specific neutralising antibodies using the GenScript® cPass surrogate virus neutralization test (sVNT) for both wild-type and Omicron variant. Neutralising antibody response will be reported as percentage (%) inhibition of receptor binding domain-angiotensin-converting enzyme 2 (RBD-ACE2) binding relative to a positive control.
Time Frame: Baseline (pre booster), 28 days-, 6- and 12-months post booster vaccination
Reporting Status: Not Posted

8. Secondary Outcome: SARS-CoV-2 Specific Neutralising Antibodies at Baseline (Pre Booster), 28 Days-, 6- and 12-months Post Booster Vaccination Measured by SARS-CoV-2 Microneutralisation Assay
Description: A subset of samples (20%) from all four timepoints will be assessed using a SARS-CoV-2 microneutralisation assay to both the wild type (vaccine) strain and for two SARS-CoV-2 Variants of concern. Neutralizing antibody will be reported as endpoint titre.
Time Frame: Baseline (pre booster), 28 days-, 6- and 12-months post booster vaccination
Reporting Status: Not Posted

9. Secondary Outcome: Interferon Gamma (IFNγ) Concentrations in International Units (IU)/mL
Description: Applicable to the subset participants with additional blood collection. Interferon gamma (IFNγ) concentrations as a measurement of cellular immunity will be assessed on a subset of the participants from each group. QuantiFERON Human IFN-γ SARS-CoV-2 (Qiagen) will be used to stimulate IFN-γ production in peripheral blood mononuclear cells (PBMCs) and then IFN-γ production will be measured using ELISA (enzyme-linked immunosorbent assay). Data will be presented as GMC and 95% CI.
Time Frame: Baseline (pre booster), 28 days-, 6- and 12-months post booster vaccination
Reporting Status: Not Posted

10. Secondary Outcome: Number of IFNγ Producing Cells/Million PBMCs
Description: Applicable to the subset participants with additional blood collection. IFNγ producing cells as a measurement of cellular immunity will be assessed on a subset of the participants (40%) from each group. IFN-γ Enzyme-Linked ImmunoSpot (Elispot) assay will be performed on isolated peripheral blood mononuclear cells (PBMCs). Data will be reported as number of IFNγ producing cells/million and presented using means and 95% CI.
Time Frame: Baseline (pre booster), 28 days-, 6- and 12-months post booster vaccination
Reporting Status: Not Posted

11. Secondary Outcome: Frequency of Cytokine-expressing T Cells
Description: Frequency of cytokine-expressing T cells will be assessed on a subset of participants (40%) using flow cytometry (intracellular staining) on PBMCs samples. Data will be reported as frequency (%) of cytokine-expressing T cells presented as means and 95% CI.
Time Frame: Assessed at 4 time-points (baseline, 28 days, 6 months, and 12 months)
Reporting Status: Not Posted

12. Secondary Outcome: Cellular Immunity: Multiplex Cytokine Assays - Reported as Cytokine Concentrations in pg/ml and Presented as GMC and 95% CI
Description: Cytokine concentrations following PBMCs stimulation will be assessed on a subset of participants (40%) using multiplex cytokine assays.Data will be reported as cytokine concentrations in pg/ml and presented as GMC and 95% CI.IFN-γ Elispot, intracellular cytokine assays (flow cytometry) and multiplex cytokine assays will be performed on isolated PBMCs.
Time Frame: Baseline (pre booster), 28 days-, 6- and 12-months post booster vaccination
Reporting Status: Not Posted

13. Secondary Outcome: Incidence of Unsolicited Adverse Events (AE)
Description: All unsolicited AE will be collected for 28 days post booster vaccination. Data will be presented as proportion of participants who report unsolicited AE.
Time Frame: 28 days-post booster vaccination
Population: The reactogenicity and safety analysis populations included all randomised participants who received a study vaccine, according to the vaccine received
Measure: Count of Participants; unit: Participants
Groups:
- Standard Pfizer-BioNTech Booster Group- AstraZeneca: Previously received two doses of AstraZeneca as primary COVID-19 vaccine
  Tozinameran - Standard Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 30 µg in 0.3 ml. Liquid for injection. Single dose.
- Fractional Pfizer-BioNTech Booster Group- AstraZeneca: Previously received two doses of AstraZeneca as primary COVID-19 vaccine
  .
  Tozinameran - Fractional Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.15 ml. Liquid for injection. Single dose.
- Standard Pfizer-BioNTech Booster Group- Sinopharm: Previously received two doses of Sinopharm as primary COVID-19 vaccine
  Tozinameran - Standard Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 30 µg in 0.3 ml. Liquid for injection. Single dose.
- Fractional Pfizer-BioNTech Booster Group- Sinopharm: Previously received two doses of Sinopharm as primary COVID-19 vaccine
  .
  Tozinameran - Fractional Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.15 ml. Liquid for injection. Single dose.
- Standard Pfizer-BioNTech Booster Group-Sputnik: Previously received two doses of Sputnik as primary COVID-19 vaccine
  Tozinameran - Standard Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 30 µg in 0.3 ml. Liquid for injection. Single dose.
- Fractional Pfizer-BioNTech Booster Group- Sputnik: Previously received two doses of Sputnik as primary COVID-19 vaccine
  .
  Tozinameran - Fractional Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.15 ml. Liquid for injection. Single dose.
Arm/Group | Standard Pfizer-BioNTech Booster Group- AstraZeneca | Fractional Pfizer-BioNTech Booster Group- AstraZeneca | Standard Pfizer-BioNTech Booster Group- Sinopharm | Fractional Pfizer-BioNTech Booster Group- Sinopharm | Standard Pfizer-BioNTech Booster Group-Sputnik | Fractional Pfizer-BioNTech Booster Group- Sputnik
Number analyzed (Participants) | 65 | 64 | 200 | 199 | 34 | 36
Participants | 5 | 9 | 12 | 7 | 5 | 5

14. Secondary Outcome: Incidence of Medically Attended Adverse Events
Description: All participants with medically attended AE will be collected for 3 months post booster vaccination. Data will be presented as proportion of participants who report unsolicited AE.
Time Frame: 3 months post booster vaccination
Reporting Status: Not Posted

15. Secondary Outcome: Incidence of Serious Adverse Events (SAE)
Description: SAE will be collected throughout the follow-up period of 12 months post booster vaccination. Data will be presented as a proportion of participants who report unsolicited SAE.
Time Frame: 12 months post booster vaccination
Reporting Status: Not Posted

16. Secondary Outcome: Incidence of PCR Confirmed COVID-19 Infection
Description: Confirmed COVID-19 infections will be documented throughout the follow-up period, by clinical severity.
Time Frame: Up to 12 months post booster vaccination
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Solicited local and systemic adverse events (AEs) were collected from the participants 7 days post-vaccination Unsolicited AEs up to 28 days following vaccination observed by the Investigator or reported by the participant, whether or not attributed to study medication, were also collected. Serious adverse events (SAE's) will be followed up for the duration of the trial up to 24 months.
Groups:
- Fractional Pfizer-BioNTech Booster Group- AstraZeneca: Previously received two doses of AstraZeneca as primary COVID-19 vaccine.
  Tozinameran - Fractional Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.15 ml. Liquid for injection. Single dose.
- Fractional Pfizer-BioNTech Booster Group- Sinopharm: Previously received two doses of Sinopharm as primary COVID-19 vaccine.
  Tozinameran - Fractional Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.15 ml. Liquid for injection. Single dose.
- Standard Pfizer-BioNTech Booster Group- Sputnik: Previously received two doses of Sputnik as primary COVID-19 vaccine
  Tozinameran - Standard Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 30 µg in 0.3 ml. Liquid for injection. Single dose.
- Fractional Pfizer-BioNTech Booster Group- Sputnik: Previously received two doses of Sputnik as primary COVID-19 vaccine.
  Tozinameran - Fractional Dose: Tozinameran is a single-stranded, 5'-capped messenger RNA (mRNA) produced using a cellfree in vitro transcription from the corresponding DNA templates, encoding the viral spike (S) protein of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
  Dose - 15 µg in 0.15 ml. Liquid for injection. Single dose.
Arm/Group | Standard Pfizer-BioNTech Booster Group- AstraZeneca | Fractional Pfizer-BioNTech Booster Group- AstraZeneca | Standard Pfizer-BioNTech Booster Group- Sinopharm | Fractional Pfizer-BioNTech Booster Group- Sinopharm | Standard Pfizer-BioNTech Booster Group- Sputnik | Fractional Pfizer-BioNTech Booster Group- Sputnik
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65 | 0/201 | 0/200 | 0/34 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/65 | 2/65 | 2/201 | 0/200 | 1/34 | 0/36
Other Adverse Events (participants affected / at risk) | 5/65 | 7/65 | 10/201 | 7/200 | 5/34 | 5/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Pfizer-BioNTech Booster Group- AstraZeneca (N=65) | Fractional Pfizer-BioNTech Booster Group- AstraZeneca (N=65) | Standard Pfizer-BioNTech Booster Group- Sinopharm (N=201) | Fractional Pfizer-BioNTech Booster Group- Sinopharm (N=200) | Standard Pfizer-BioNTech Booster Group- Sputnik (N=34) | Fractional Pfizer-BioNTech Booster Group- Sputnik (N=36)
Hepatobiliary (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Pfizer-BioNTech Booster Group- AstraZeneca (N=65) | Fractional Pfizer-BioNTech Booster Group- AstraZeneca (N=65) | Standard Pfizer-BioNTech Booster Group- Sinopharm (N=201) | Fractional Pfizer-BioNTech Booster Group- Sinopharm (N=200) | Standard Pfizer-BioNTech Booster Group- Sputnik (N=34) | Fractional Pfizer-BioNTech Booster Group- Sputnik (N=36)
Abdominal cramps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Allergy to chemicals (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Natural menopause (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/65/NCT05265065/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-23): https://cdn.clinicaltrials.gov/large-docs/65/NCT05265065/SAP_002.pdf